CLINICAL TRIAL: NCT02739971
Title: Dietary Reduction of Advanced Glycation End Products to Prevent Cognitive Decline in Elderly Diabetics - a Randomized Pilot Trial
Brief Title: Dietary Reduction of AGEs to Prevent Cognitive Decline in Elderly Diabetics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Hebrew University of Jerusalem (Other)
Responsible Party: Principal Investigator, Dr. Ithamar Ganmore, Principle investigator, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SHEBA-15-2206-IG-CTIL
Record Dates: First submitted 2016-04-05; First posted 2016-04-15 (Estimated); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Cognitive Decline; Aging; Type 2 Diabetes
MeSH Terms: conditions — Cognitive Dysfunction; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: A randomized pilot trial
Who Masked: Outcomes Assessor
Masking Description: The participants and study dietitian can not be blind to the assigned dietary intervention. However, the clinical testing and all data analysis are carried out blind to the intervention.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low AGEs diet (Active Comparator): Participants randomized to this arm will receive active instruction on reducing dietary AGEs intake, in addition to standard of care dietary guidance for type 2 diabetes.
  Interventions: Behavioral: Low AGEs diet; Behavioral: Standard of care dietary guidance for Type 2 diabetes
- Standard of care dietary guidance (Placebo Comparator): Participants randomized to this arm will only recieve standard of care dietary guidance for type 2 diabetes.
  Interventions: Behavioral: Standard of care dietary guidance for Type 2 diabetes

INTERVENTIONS:
Behavioral: Low AGEs diet — Oral and written instructions on how to reduce AGEs in diet, mainly by changing cooking methods in addition to standard of care dietary guidance for type 2 diabetes
  Arms: Low AGEs diet
Behavioral: Standard of care dietary guidance for Type 2 diabetes — Oral and written instructions for standard of care dietary guidance for type 2 diabetes

SUMMARY:
Basic science and observational human studies suggest that high conentrations of circulating Advanced Glycation End-products (AGEs) may promote cognitive decline in older adults. The purpose of this pilot study is to test the methodology and feasibility of a dietary intervention to lower AGEs in elderly diabetics in order to lay the foundations for a future fully powered randomized clinical trial (RCT).To this end, the present study is focused on recruitment strategies, adherence to an innovative intervention in older adults and study methods. An exploratory aim will be the effect of the intervention on cognition and cerebral blood flow in order to obtain necessary data to estimate effect-size for a future fully-powered RCT.

ELIGIBILITY:
* Above the age 65
* T2D diagnosis
* no dementia (i.e MCI or cognitively normal )
* Not receiving cholinesterase inhibitors
* No other neurological (e.g. stroke, Parkinson's disease) or psychiatric conditions (e.g. schizophrenia, depression) that may affect cognition
* Dietary AGE levels > 13kU
* Not participating in another clinical trial
* An informant that is willing to actively support the participant throughout the study

Exclusion Criteria:

* Dementia
* Stroke
* Other major neuropsychiatric condition that might affect cognition

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 75 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in AGEs markers in serum (carboxymethyl lysine, CML and Methylglyoxal ,MG ) at 6 months | 6 months
  Blood draws before and at the end of the intervention

SECONDARY OUTCOMES:
recruiting rate assessment | 2 years of total recruitment
  calculate the eligible subjects from those attended screening visit
retention rate to the diet | 6 months
  to report the retention rate

OTHER OUTCOMES:
The influence of AGE reduction on cognition | 6 months
  Changes in cognition using a Z score of global and domain specific (language, attention, memory ) cognition following 6 months of AGEs reduction compared to standard of care (this is an exploratory aim since this is a pilot study)
The influence of AGE reduction on cerebral blood flow-measured with arterial spin labeling MRI (ASL-MRI) | 6 months
  changes in cerebral blood flow measured with ASL MRI following 6 months of AGEs reduction compared to standard of care ( this is an exploratory aim since this is a pilot study)
Change in microbial diversity and composition of fecal microbiome following AGE reduction in diet | 6 months
  microbiota composition will be analyzed (eg. the amount and relative proportions of major bacterial genus and species Bifidobacterium, Bacteroides, Lactobaillus, Enterobacteria, Eubacteria,etc. using 16S rRNA profiling ) before and after intervention of AGEs reduction and changes will compared to standard of care arm. This is a descriptive exploratory outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Michal Schnaider Beeri, PhD, Principal Investigator — The Joseph Sagol Neuroscience Center; Aron M Troen, DPhil, Principal Investigator — Hebrew University of Jerusalem; Ramit Ravona Springer, MD, Study Director — The Joseph Sagol Neuroscience Center
Locations (1):
- Joseph Sagol Neuroscience center, Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Uribarri J, Woodruff S, Goodman S, Cai W, Chen X, Pyzik R, Yong A, Striker GE, Vlassara H. Advanced glycation end products in foods and a practical guide to their reduction in the diet. J Am Diet Assoc. 2010 Jun;110(6):911-16.e12. doi: 10.1016/j.jada.2010.03.018. PMID 20497781
- [Background] Cai W, Uribarri J, Zhu L, Chen X, Swamy S, Zhao Z, Grosjean F, Simonaro C, Kuchel GA, Schnaider-Beeri M, Woodward M, Striker GE, Vlassara H. Oral glycotoxins are a modifiable cause of dementia and the metabolic syndrome in mice and humans. Proc Natl Acad Sci U S A. 2014 Apr 1;111(13):4940-5. doi: 10.1073/pnas.1316013111. Epub 2014 Feb 24. PMID 24567379
- [Background] Lubitz I, Ricny J, Atrakchi-Baranes D, Shemesh C, Kravitz E, Liraz-Zaltsman S, Maksin-Matveev A, Cooper I, Leibowitz A, Uribarri J, Schmeidler J, Cai W, Kristofikova Z, Ripova D, LeRoith D, Schnaider-Beeri M. High dietary advanced glycation end products are associated with poorer spatial learning and accelerated Abeta deposition in an Alzheimer mouse model. Aging Cell. 2016 Apr;15(2):309-16. doi: 10.1111/acel.12436. Epub 2016 Jan 19. PMID 26781037
- [Background] Uribarri J, Cai W, Ramdas M, Goodman S, Pyzik R, Chen X, Zhu L, Striker GE, Vlassara H. Restriction of advanced glycation end products improves insulin resistance in human type 2 diabetes: potential role of AGER1 and SIRT1. Diabetes Care. 2011 Jul;34(7):1610-6. doi: 10.2337/dc11-0091. PMID 21709297
- [Background] Ravona-Springer R, Luo X, Schmeidler J, Wysocki M, Lesser G, Rapp M, Dahlman K, Grossman H, Haroutunian V, Schnaider Beeri M. Diabetes is associated with increased rate of cognitive decline in questionably demented elderly. Dement Geriatr Cogn Disord. 2010;29(1):68-74. doi: 10.1159/000265552. Epub 2010 Jan 30. PMID 20130405
- [Background] Luchsinger JA, Reitz C, Patel B, Tang MX, Manly JJ, Mayeux R. Relation of diabetes to mild cognitive impairment. Arch Neurol. 2007 Apr;64(4):570-5. doi: 10.1001/archneur.64.4.570. PMID 17420320
- [Background] Beeri MS, Moshier E, Schmeidler J, Godbold J, Uribarri J, Reddy S, Sano M, Grossman HT, Cai W, Vlassara H, Silverman JM. Serum concentration of an inflammatory glycotoxin, methylglyoxal, is associated with increased cognitive decline in elderly individuals. Mech Ageing Dev. 2011 Nov-Dec;132(11-12):583-7. doi: 10.1016/j.mad.2011.10.007. Epub 2011 Nov 3. PMID 22079406
- [Background] West RK, Moshier E, Lubitz I, Schmeidler J, Godbold J, Cai W, Uribarri J, Vlassara H, Silverman JM, Beeri MS. Dietary advanced glycation end products are associated with decline in memory in young elderly. Mech Ageing Dev. 2014 Sep;140:10-2. doi: 10.1016/j.mad.2014.07.001. Epub 2014 Jul 15. PMID 25037023
- [Derived] Lotan R, Ganmore I, Livny A, Shelly S, Zacharia M, Uribarri J, Beisswenger P, Cai W, Schnaider Beeri M, Troen AM. Design and Feasibility of a Randomized Controlled Pilot Trial to Reduce Exposure and Cognitive Risk Associated With Advanced Glycation End Products in Older Adults With Type 2 Diabetes. Front Nutr. 2021 Feb 15;8:614149. doi: 10.3389/fnut.2021.614149. eCollection 2021. PMID 33659267
- [Derived] Lotan R, Ganmore I, Shelly S, Zacharia M, Uribarri J, Beisswenger P, Cai W, Troen AM, Schnaider Beeri M. Long Term Dietary Restriction of Advanced Glycation End-Products (AGEs) in Older Adults with Type 2 Diabetes Is Feasible and Efficacious-Results from a Pilot RCT. Nutrients. 2020 Oct 15;12(10):3143. doi: 10.3390/nu12103143. PMID 33076217